CLINICAL TRIAL: NCT04760405
Title: The TOTOM Trial: Tai Chi to Optimize Transplant Outcomes for Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011190017
Record Dates: First submitted 2021-01-15; First posted 2021-02-18 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma; Stem Cell Transplant Complications
Keywords: Multiple Myeloma; Stem cell transplant; Autologous stem cell transplantation; ASCT; Tai Chi
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi Easy Intervention (Experimental): Tai Chi Easy: TCE is a standardized protocol used in several prior studies. TCE has been manualized and has a formal training program for instructors. The protocol is taught as a series of repeated and simple-to-learn movements. Patients will receive two 30-minute small group training sessions (Via Zoom) within 7 days of their scheduled transplant. After the training has been completed the participant will be provided with written (via manual) and electronic (DVD, MP3 file download) materials to continue with self-direct practice throughout the duration of the study.
  Interventions: Other: Tai Chi Easy

INTERVENTIONS:
Other: Tai Chi Easy — Patients will receive two 30-minute small group training sessions (Via Zoom) within 7 days of their scheduled transplant. After the training has been completed the participant will be provided with written (via manual) and electronic (DVD, MP3 file download) materials to continue with self-direct practice throughout the duration of the study.

SUMMARY:
The current proposal aims to test the feasibility of immune function analysis for Tai Chi Easy (TCE) intervention in multiple myeloma (MM) patients undergoing autologous stem cell transplantation (ASCT) with concurrent exploration of health related quality of life (HRQOL).

DETAILED DESCRIPTION:
The current proposal aims to test the feasibility of immune function analysis for TCE intervention in MM patients undergoing ASCT with concurrent exploration of HRQOL. The data obtained from this trial will provide supporting data for a future randomized clinical trial evaluating the impact of TCE on immune function (incidence of ASCT related infectious complications, natural killer cell phenotype and activity, and myeloma remission rate (clonal plasma cell % at day 100, minimal residual disease (MRD)), with the evaluation of efficacy on improving HRQOL during ASCT. Successful completion of this CROC project will provide necessary data to support future grant applications, in particular the feasibility of immunoassay evaluation of MM patients undergoing ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Myeloma planned to undergo bone marrow transplant
2. 18 years or older
3. English speaking
4. General proficiency to read/write in English
5. Able to attend TCE training session per study protocol
6. ECOG performance status 0-1
7. Able to return to study center for routine post-transplant follow up (approximately Day 30 and Day 100)

Exclusion Criteria:

1. Currently performs Tai Chi, QiQong, or Yoga at least once weekly or more
2. Syncopal event in prior 60 days
3. Concurrent major depressive disorder or anxiety disorder (DSMIV) as determined by treating provider
4. Chronic dizziness or vestibular disorders
5. History of recurrent falls (>2 in the prior year)
6. Grade 3 or greater neuropathy
7. Grade 3 or greater spinal fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Determine natural killer cell phenotype | Baseline
  Determine natural killer (NK) phenotype through peripheral blood analysis
Determine natural killer cell phenotype | Day 14
  Determine natural killer (NK) phenotype through peripheral blood analysis
Determine natural killer cell phenotype | Day 30
  Determine natural killer (NK) phenotype through peripheral blood analysis
Determine natural killer cell phenotype | Day 100
  Determine natural killer (NK) phenotype through peripheral blood analysis
Determine NK cell activity | At baseline
  Determine NK cell activity through peripheral blood analysis
Determine NK cell activity | Day 14
  Determine NK cell activity through peripheral blood analysis
Determine NK cell activity | Day 30
  Determine NK cell activity through peripheral blood analysis
Determine NK cell activity | Day 100
  Determine NK cell activity through peripheral blood analysis
Determine immune function | At baseline
  Determine immune function through peripheral blood analysis of immune factors
Determine immune function | Day 14
  Determine immune function through peripheral blood analysis of immune factors
Determine immune function | Day 30
  Determine immune function through peripheral blood analysis of immune factors
Determine immune function | Day 100
  Determine immune function through peripheral blood analysis of immune factors

CONTACTS AND LOCATIONS:
Overall Officials: Krisstina Gowin, DO, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Mayo Clinic, Jacksonville, Florida